CLINICAL TRIAL: NCT07052526
Title: Evaluation of Hydrophilic and Hydrophobic Sealants' Retention, Caries Prevention, Microleakage, and Fluoride Release in Partially Erupted First Permanent Molars:A Randomized Controlled Clinical Trial
Brief Title: Comparative Evaluation of Hydrophilic and Hydrophobic Sealants in Partially Erupted First Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Mohamed, Assisstant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MU-DPH-Heba2025
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Dental Caries
Keywords: Hydrophilic sealant;; Fluoride; Microleakage; Caries; Retention
MeSH Terms: conditions — Dental Caries | interventions — Secondary Prevention

STUDY DESIGN:
Intervention Model Description: A total of 150 children aged 5-7 will be randomly assigned to three equal groups of 50 participants each
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Helioseal Fplus (Experimental): Participants in this arm will receive the Helioseal F Plus resin-based sealant, applied to occlusal surfaces of permanent molars. The sealant will be applied according to the manufacturer's
  Interventions: Other: Prevention
- 1 - Hydrophilic Sealant (Embrace WetBond) (Experimental): Participants will receive Embrace WetBond sealant, a moisture-tolerant resin sealant applied to slightly moist occlusal surfaces. The sealant is light-cured for 20 seconds
  Interventions: Other: Prevention of caries
- Denu seal (Experimental): Participants in this arm will receive Denuseal, a fluoride-releasing sealant, applied to occlusal surfaces of permanent molars under dry conditions. The sealant will be light-cured for 20 seconds.
  Interventions: Other: Prevention therapy

INTERVENTIONS:
Other: Prevention — Conventional Hydrophobic Sealant (Helioseal F - Control) will be used as a positive control; applied to partially erupted molars with and without bonding in a split-mouth design.
  Other Names: Helioseal-F plus
  Arms: Helioseal Fplus
Other: Prevention of caries — Embrace WetBond sealant will be applied to partially erupted first permanent molars using a split-mouth design with and without bonding agent.
  Other Names: Hydrophilic Embrace-Wetbond
  Arms: 1 - Hydrophilic Sealant (Embrace WetBond)
Other: Prevention therapy — DENU Seal applied using a split-mouth design to evaluate bonding and non-bonding application outcomes from retention and caries prevention
  Other Names: Denuseal
  Arms: Denu seal

SUMMARY:
This randomized controlled clinical trial aims to evaluate and compare the retention, caries prevention, microleakage, and fluoride release of three types of pit and fissure sealants-hydrophilic, nanofilled hydrophobic, and conventional hydrophobic-applied to partially erupted first permanent molars in children aged 5 to 7 years. The study uses a split-mouth design and includes both clinical and laboratory evaluations over an 18-month period. Outcomes will assess sealant effectiveness with and without the use of a bonding agent.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial designed to evaluate and compare the effectiveness of three types of pit and fissure sealants-hydrophilic (Embrace WetBond), nanofilled hydrophobic (DENU Seal), and conventional hydrophobic (Helioseal F)-when applied to partially erupted first permanent molars in children aged 5 to 7 years. The study aims to assess the sealants' clinical retention, their ability to prevent dental caries, microleakage, sealant penetration depth, and fluoride release.

A total of 150 children will be randomly assigned to three equal groups of 50 participants each. A split-mouth design will be used: in each group, sealants will be applied with and without bonding agents on opposite sides of the upper or lower arch, allowing intra-subject comparisons. Clinical evaluations will be conducted at 3, 6, 12, and 18 months to assess sealant retention and caries incidence using the modified Color, Coverage, Caries (CCC) Sealant Evaluation System.

In addition to the clinical phase, a laboratory phase will be conducted using extracted human premolars. This phase will evaluate microleakage and sealant penetration under a stereomicroscope following dye penetration techniques. Fluoride release will be measured at specified time intervals (1, 7, 14, 21, and 28 days) using an ion-selective electrode in artificial saliva conditions maintained at 37°C.

The primary outcomes include sealant retention and caries incidence. Secondary outcomes focus on the degree of microleakage, sealant penetration, and fluoride release. The trial will help determine whether moisture-tolerant sealants offer superior clinical and preventive benefits over traditional hydrophobic materials, particularly in situations where ideal isolation is difficult, such as with partially erupted teeth in young children.

The study will be conducted at the Pediatric Dentistry Clinic, Faculty of Dentistry, Mansoura University, and is expected to generate evidence that could improve clinical decision-making in preventive pediatric dentistry.

ELIGIBILITY:
-

Inclusion Criteria:

* Cooperative children (Frankl Scale 3)
* good oral hygiene (OHI-S Index),
* 2 partially erupted 1st molars

Exclusion Criteria:

* Cavitated caries
* fluorosis
* hypoplasia
* restored teeth

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — All
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Retention | 18 months
  retention is evaluated using CCC Index (Color, Coverage, and Caries)
  This scale is used to assess sealant retention and caries status during follow-up evaluations.
  Score Description Retention Caries Status Interpretation
  0 Sealant completely retained no caries Full retention Best outcome
  1. Partial sealant loss no caries Partial loss Acceptable
  2. Sealant completely lost no caries Total loss Less ideal
  3. Sealant partially or totally lost caries present Partial or total loss Worst outcome
Caries | 18 months
  Caries Incidence: 3, 6, 12, 18 months, t each recall (3, 6, 12 months), evaluate each sealed tooth using the CCC score:
  If the sealant is completely intact and no caries is visible → score = 0
  If the sealant is partially gone but no decay → score = 1
  If sealant is lost but still no decay → score = 2
  If sealant is lost/partial and there is decay → score = 3

SECONDARY OUTCOMES:
Microleakage | 3 months
  Microleakage Assessment (lab) - dye penetration . Score Description Microleakage Depth Interpretation
  0 No dye penetration 0% of fissure depth Best outcome
  1. Dye penetrates into enamel only <50% of enamel Good
  2. Dye penetrates to dentino-enamel junction (DEJ) Reaches DEJ, no dentin Borderline
  3. Dye penetrates into dentin Past DEJ into dentin Worst outcome
  Minimum score: 0 = no leakage
  Maximum score: 3 = extensive leakage
  Higher score = worse outcome
Fluoride release | 2months
  Fluoride Release - spectrophotometer (1, 7, 14, 21, 28 days) Fluoride Release Scoring System (Modified Scale for Clinical Correlation)
  Because fluoride release is continuous and measured in ppm or µg/cm²/day, we can categorize release levels into scores for easier interpretation.
  Score Fluoride Release Level Typical Range Interpretation
  0 High, sustained release >2 ppm after 1 week Best outcome
  1. Moderate release 1-2 ppm after 1 week Good
  2. Low release 0.5-1 ppm after 1 week Weak effect
  3. Negligible release <0.5 ppm after 1 week Ineffective

CONTACTS AND LOCATIONS:
Overall Officials: Dr rabaa MAHMOUD ABOU Bakr, Professor, Principal Investigator — Mansoura University - Pediatric Dentistry Clinic
Locations (1):
- Facility of Dentistry،Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request for academic use.
Time Frame: 2 years
Access Criteria: Researcher
URL: https://heba.mohamed@mans.edu.eg

REFERENCES:
- See also: This randomized controlled trial compared hydrophilic (UltraSeal XT Hydro) and hydrophobic (Helioseal-F) resin-based sealants in uncooperative childre in aged 6-9 years. Using a split-mouth design, sealants were applied to 49 pairs of molars and assessed — https://pubmed.ncbi.nlm.nih.gov/39087225/
- See also: In-vitro studies on pit and fissure sealants often involve measuring fluoride ion release to assess their potential anticariogenic effects. Fluoride release is typically measured using a fluoride ion-selective electrode and an ion analyzer. Different typ — https://www.jstage.jst.go.jp/article/tdcpublication/45/3/45_3_173/_pdf